CLINICAL TRIAL: NCT02937636
Title: A Clinical Study Investigating the Gingivitis Efficacy of a Stannous Fluoride Dentifrice in a Chinese Population.
Brief Title: To Investigate the Gingivitis Efficacy of a Stannous Fluoride Dentifrice in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207014
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): Participants will apply a full strip of dentifrice to cover the head of the toothbrush provided and brush their teeth with the assigned dentifrice twice daily (morning and evening) for one timed minute following their normal routine.
  Interventions: Other: Stannous fluoride
- Reference Product (Active Comparator): Participants will apply a full strip of dentifrice to cover the head of the toothbrush provided and brush their teeth with the assigned dentifrice twice daily (morning and evening) for one timed minute following their normal routine.
  Interventions: Other: Sodium monofluorophosphate

INTERVENTIONS:
Other: Stannous fluoride — Experimental dentifrice containing 0.454% w/w stannous fluoride & 0.0721% w/w sodium fluoride containing1450 parts per million (ppm) fluoride
  Arms: Test Product
Other: Sodium monofluorophosphate — Dentifrice containing 0.14% w/w sodium monofluorophosphate containing1400 ppm fluoride
  Arms: Reference Product

SUMMARY:
This single-centre, examiner-blind, randomized, stratified, two-treatment, parallel group clinical study will evaluate the efficacy of a 0.454% w/w stannous fluoride dentifrice compared to a reference dentifrice to control gingivitis (gingival bleeding and visual signs of gingival inflammation) in dentally and periodontally healthy adult volunteers over 12 weeks use in a Chinese population.

DETAILED DESCRIPTION:
This clinical study will be carried out in healthy adult volunteers with moderate gingivitis. Treatment effect will be determined by evaluating the efficacy, in a Chinese population, of a dentifrice containing 0.454% w/w stannous fluoride to control gingivitis and supra-gingival plaque following 6 and 12 weeks twice daily brushing, compared to a fluoride control dentifrice. During the 12 week treatment period, participant will brush with their allocated study product twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged 18 to 65 years.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon oral examination, absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* A minimum of 20 natural teeth (all teeth; incisors, canines, pre-molars & molars), and a minimum of 40 gradable surfaces for MGI, BI and PI. A scorable surface is defined as a surface that has 50% of the surface gradable for each clinical index. Third molars, orthodontically banded/bonded, fully crowned or extensively restored or grossly carious teeth are not included in the tooth count, moderate gingivitis present at the screening visit (in the opinion of the clinical examiner from a gross visual examination) and mean whole mouth MGI between 1.75 and 2.30 and a mean overall PI score >1.5 at Baseline visit.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Screening: Currently taking antibiotics or requiring antibiotic use prior to dental prophylaxis or other dental procedures, currently taking an anti-inflammatory medication or traditional Chinese medicines (TCM) which, in the opinion of the Investigator, could affect gingival condition, currently taking a systemic medication which, in the opinion of the Investigator, could affect gingival condition (e.g. calcium channel blockers, or aspirin therapy).
* Baseline (Visit 2): Has taken, or currently taking, antibiotics in the previous 14 days, or an anti-inflammatory medication or a systemic medication days (e.g. calcium channel blockers, or aspirin therapy) which, in the opinion of the Investigator, could affect gingival condition in the previous 14 days.
* Have current active caries or periodontitis that may, in the opinion of the investigator, compromise the study or the oral health of the participants if they participate in the study, restorations in a poor state of repair, partial dentures or orthodontic appliances, teeth bleaching within 12 weeks of screening and use of a chlorhexidine mouthwash currently, or within 14 days of baseline.
* Participation in another clinical study or receipt of an investigational drug or investigational oral care product within 30 days of Baseline (Visit 2) and previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family and employed by any dentifrice manufacturer or their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in China.
Pre-assignment Details: A total of 343 participates were screened, out of which 128 participants were randomized in the study. 215 participants were not randomized as 186 participants did not meet study criteria, 5 participants withdrew consent and 24 were not randomized for other reasons (not specified).
Groups:
- Test Product: Participants applied a full strip of dentifrice containing 0.454% weight by weight (w/w) stannous fluoride and 0.0721% w/w sodium fluoride containing 1450 parts per million (ppm) fluoride to cover the head of the toothbrush provided and brush their teeth with the assigned dentifrice twice daily (morning and evening) for one timed minute following their normal routine.
- Reference Product: Participants applied a full strip of dentifrice containing 0.14% w/w sodium monofluorophosphate (1400 ppm fluoride) to cover the head of the toothbrush provided and brush their teeth with the assigned dentifrice twice daily (morning and evening) for one timed minute following their normal routine.
Period: Overall Study
Arm/Group | Test Product | Reference Product
Started | 63 | 65
Completed | 60 | 63
Not Completed | 3 | 2
Not completed — Other (Not specified) | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population (n=128) included all participants who were randomized and received at least one dose of study products.
Groups:
- Test Product: Participants applied a full strip of dentifrice containing 0.454% w/w stannous fluoride and 0.0721% w/w sodium fluoride containing 1450 ppm fluoride to cover the head of the toothbrush provided and brush their teeth with the assigned dentifrice twice daily (morning and evening) for one timed minute following their normal routine.
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Customized [Mean (Standard Deviation); unit: Years] | 40.8 (10.20) | 42.9 (10.04) | 41.9 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 63 | 65 | 128
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Stratification n (%) [Count of Participants; unit: Participants]
  Male, Smoker, Baseline MGI <= 2.00 | 0 | 0 | 0
  Male, Smoker, Baseline MGI > 2.00 | 1 | 1 | 2
  Male, non-smoker, Baseline MGI <= 2.00 | 0 | 0 | 0
  Male, non-smoker, Baseline MGI > 2.00 | 11 | 12 | 23
  Female, Smoker, Baseline MGI <= 2.00 | 0 | 0 | 0
  Female, Smoker, Baseline MGI > 2.00 | 0 | 0 | 0
  Female, non-smoker, Baseline MGI <= 2.00 | 4 | 3 | 7
  Female, non-smoker, Baseline MGI > 2.00 | 47 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: Mean Bleeding Index (BI)
Description: The BI was performed by a single examiner using a color coded periodontal probe. The probe was inserted approximately 1 mm into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system to be used is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed. This measure will be analyzed and summarized over all sites.
Time Frame: At Week 12
Population: The intent to treat (ITT) (n=128) population is defined as those participants who were randomized, received at least one dose of study product and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 63 | 65
Score on Scale | 0.07 (0.059) | 0.15 (0.128)
Statistical Analysis 1: Comparison: Reference Product; Test type: Other; p < .0001, ANCOVA; From ANCOVA with treatment, gender, smoking status and baseline MGI stratification as factors and baseline as covariate; Least square (LS) mean difference = -0.09, 95% CI 2-sided [-0.12 to -0.07] — Difference is the first named treatment minus second named treatment such that a negative difference favors the first named treatment

2. Secondary Outcome: Number of Bleeding Sites
Description: Number of bleeding sites were measured as BI via a single examiner using a color coded periodontal probe. The probe was gently inserted approximately 1 millimeter (mm) into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system used to measure bleeding sites is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed. A bleeding site was considered as a BI score of 1 or 2.
Time Frame: At Week 12
Population: The ITT (n=128) population is defined as those participants who were randomized, received at least one dose of study product and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Number of bleeding sites
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 63 | 65
Number of bleeding sites | 10.37 (8.499) | 20.92 (15.881)

3. Secondary Outcome: Mean Modified Gingival Index (MGI)
Description: The MGI was assessed on facial and lingual surfaces at two sites on each tooth (papillae and margin).The scoring of MGI was performed by a single examiner. The MGI scoring system is as follows:0=absence of inflammation;1=mild inflammation; slight change in color, little change in color; little change in texture of any portion of the marginal or papillary gingival unit;2=mild inflammation; criteria as above but involving the entire marginal or papillar gingival units;3=moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit;4=severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration.
Time Frame: At Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score On Scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 63 | 65
Score On Scale | 1.62 (0.211) | 1.89 (0.198)

4. Secondary Outcome: Mean Plaque Index (PI) (Overall and Interproximal)
Description: The dental examiner used the PI to assess plaque on all gradable teeth. The plaque was first disclosed using a dye solution. Participants then rinsed with disclosing solution according to instructions. Plaque was assessed with each tooth being divided into 6 areas including the mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces. Disclosed plaque was scored as follows: 0= No plaque; 1= Slight flecks of plaque at the cervical margin of the tooth; 2= A thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth; 3= A band of plaque wider than 1 mm but covering less than 1/3 of the crown of the tooth; 4= Plaque covering at least 1/3 but less tan 2/3 of the crown of the tooth; 5= Plaque covering 2/3 or more of the crown of the tooth.Overall PI score and interproximal PI score were calculated as the mean PI over all tooth sites and mean PI over interproximal sites (distal and mesial) respectively.
Time Frame: At Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 63 | 65
Score on Scale
  Mean Plaque Index (PI) (overall) | 1.85 (0.319) | 2.19 (0.245)
  Mean Plaque Index (PI) (interproximal) | 1.92 (0.313) | 2.24 (0.240)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Test Product | Reference Product
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/65
Other Adverse Events (participants affected / at risk) | 3/63 | 2/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=63) | Reference Product (N=65)
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT02937636/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT02937636/SAP_001.pdf